CLINICAL TRIAL: NCT00564434
Title: Postoperative Delirium in Hip Fracture Patients
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Other Study IDs: 1.2005.812
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Delirium
Keywords: delirium; pathophysiology; risk factors; pain; dementia
MeSH Terms: conditions — Delirium; Pain; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Risk factors for postoperative delirium in hip fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture
* age 65 or older

Exclusion Criteria:

* critical ill/ dying
* aphasia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with hip fracture admitted to Ulleval Hospital and Diakonhjemmet Hospital
Enrollment: 364
Dates: Start 2005-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Delirium/ no-delirium | 5 days postoperative

SECONDARY OUTCOMES:
Severity of delirium, length of delirium, complications, comorbidity, one-year mortality. | 5 days postoperative, one year

CONTACTS AND LOCATIONS:
Locations (1):
- Ullevaal Hospital, Oslo, Oslo County, Norway